CLINICAL TRIAL: NCT06411067
Title: Investigational Use of Erenumab for the Treatment of Fibromyalgia Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lapse in IRB approval
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCP.2020.0010
Record Dates: First submitted 2020-03-06; First posted 2024-05-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Chronic pain; CGRP
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — erenumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded, placebo controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Medication is drawn in unlabeled syringes by nurse. Investigators and outcomes assessors are blinded to treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): 1ml 0.9% of saline once a month in addition to the standard of care practiced at NMCP.
  Interventions: Drug: Saline
- Erenumab (Experimental): 140mg (1 ml) of Erenumab injected once a month in addition to the standard of care practiced at NMCP.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Monthly injection of erenumab for fibromyalgia
  Arms: Erenumab
Drug: Saline — Monthly injection of 0.9% saline for control
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the administration of the CGRP-receptor antagonist erenumab is effective in decreasing pain and improving quality of life in patients with FMS by comparing the difference in pain scores in Fibromyalgia Impact Questionnaire, defense and veterans Pain Rating Scale and The American College of Rheumatology 2010 Preliminary Diagnostic Criteria for Fibromyalgia score over the study period.

DETAILED DESCRIPTION:
Patients will be identified as possible participants who are referred to the Pain Management Clinic who were previously diagnosed with Fibromyalgia. At the patients' first clinic visit, explanation of the study and informed written consent will be obtained. Once consent is obtained patients will be considered enrolled in the study and will be randomized to either the experimental (erenumab) or control (saline) groups. We will plan to enroll 70 patients, 35 in each arm. Patients will undergo baseline evaluation with The American College of Rheumatology 2010 Preliminary Diagnostic Criteria for Fibromyalgia score, Defense and Veterans Pain Rating Scale (DVPRS), Fibromyalgia Impact Questionnaire, Beck Depression Inventory and CAGE-AID questionnaire. Both groups will undergo injections at t=0, t=1 month, and t=2 months, with repeat assessment of symptoms with the Fibromyalgia score, DVPRS, BDI, FIQ, at t=0, t=1 month, t= 2 months, and t=3 months.

Enrolled patients must meet the following criteria: 1) must be between the ages of 18-85; 2) a diagnosis must be made from a practicing physician; 3) existing pain for more than 3 months; 4) pain resistant to common analgesics or intolerance to common analgesic; 5) widespread pain in at least 7 of 19 areas ( as reported by the patient); 6) symptom severity scale score over five including symptoms of fatigue, awaking unrefreshed and brain fog. Exclusion criteria involve 1) positive pregnancy test, 2) drug or alcohol abuse; 3) severe depression; 4) change in CNS active medications in the previous 2 months.

Patients in both groups will undergo injections with either erenumab or saline in the clinic performed by a clinic nurse. Once enrolled, patients will be randomized by a random number generator and enrolled into either the saline or erenumab group. Because erenumab is sold as an autoinjector, the injector will be inserted into a sterile vial, and the 1mL of erenumab will be withdrawn with a tuberculin needle and then injected subcuteanously. The saline group will be injected 1mL of 0.9% saline subcutaneously. The nurse administering the injection will not be blinded, however the investigators and the subjects will be blinded to achieve double blinding. The erenumab group will be administered 140mg Subcutaneously once monthly, while the control group will be administered 1ml 0.9% saline Subcutaneously once monthly. All patients will be monitored for one hour, after the injection is administered.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of fibromyalgia made by a practicing physician between the ages of 18-85 existing pain for more than 3 months pain resistant to common analgesics or intolerance to common analgesics Active Duty service members widespread pain in at least 7 of 19 areas; as reported by the patient symptom severity scale score over five including symptoms of fatigue, awaking unrefreshed and brain fog

Exclusion Criteria:

Pregnancy ages under 18 and over 85 years of age Non Active Duty service members Anaphylactic reactions Allergy to latex Drug or alcohol abuse severe depression change in CNS active medications in the preceding 2 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Defense and Veterans Pain Rating Scale (DVPRS) | t=0, t=1 month, t=2 months, and t=3 months
  Defense and Veterans Pain Rating Scale (DVPRS)
Fibromyalgia Impact Questionnaire | t=0, t=1 month, t=2 months, and t=3 months
  Fibromyalgia Impact Questionnaire
Beck Depression Inventory | t=0, t=1 month, t=2 months, and t=3 months
  Beck Depression Inventory

SECONDARY OUTCOMES:
CAGE-AID Questionnaire | t=0, t=1 month, t=2 months, and t=3 months
  CAGE-AID Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No